CLINICAL TRIAL: NCT06373510
Title: Longitudinal Evaluation of Antibody Kinetics Following Administration of a Non-mandatory Marketed Vaccine in the General Population, Real-life Study
Brief Title: Longitudinal Evaluation of Antibody Kinetics of Vaccinated Patients With Non-mandatory Vaccine Following Administration of a Non-public Marketed Vaccine in the General Population, Real-life Study
Acronym: ELCAV
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CerbaXpert (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: ELCAV
Record Dates: First submitted 2024-04-04; First posted 2024-04-18 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Vaccination Reaction
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Observational arm (Other)
  Interventions: Biological: Blood collection

INTERVENTIONS:
Biological: Blood collection — Collection of blood before and after a non mandatory vaccination

SUMMARY:
The study would make it possible to document more explicitly the evolution of antibody titers at following a non-public vaccination over a large post-vaccination period in the French population .

Analysis of real-life data would enhance knowledge of vaccine response kinetics It would be useful to identify possible early declines requiring doses Similarly, by analyzing antibody kinetics by age, sex, and vaccination status, the would be possible to determine whether there are differences in the immune response between these different sub-groups. In addition, it would provide additional information to assess the real impact of these non-public vaccines in public health and guide vaccine policies.

ELIGIBILITY:
Inclusion Criteria:

* Subject over 18 years of age
* Subject presenting to the investigation centre as part of its usual management (prevention, screening, tracking)
* Subject who has been vaccinated and/or wishes to be vaccinated
* Subject able to understand the purpose of research that has given free and informed express consent
* Member or beneficiary of a social security scheme

Exclusion Criteria:

* Protected subject: major under guardianship, curatorship or other legal protection, deprived of liberty by decision judicial or administrative

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10000 (Estimated)
Dates: Start 2024-06-20 (Estimated); Primary Completion 2027-04-03 (Estimated); Study Completion 2027-04-03 (Estimated)

PRIMARY OUTCOMES:
Quantification of specific serum antibodies (IgM, IgG) at different times before and/or after vaccination by a reference technique such as ELISA. | 3 years
  Quantification of specific serum antibodies (IgM, IgG) at different times before and/or after vaccination by a reference technique such as ELISA.

IPD SHARING:
Plan to Share IPD: No